CLINICAL TRIAL: NCT03651674
Title: Longitudinal Effect of Electroconvulsive Therapy on Schizophrenia and Bipolar Disorder: a MRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xidian University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 81471815
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia, Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECT treatment (Active Comparator): Patients received bilateral temporal modified ECT (MECT) for three weeks,four times a week. Meanwhile, they also had antipsychotic drugs.
  Interventions: Device: ECT treatment
- Drug treatment (Sham Comparator): Patients only received antipsychotic drugs during observation period.
  Interventions: Drug: Drug treatment

INTERVENTIONS:
Device: ECT treatment — Patients had bilateral temporal modified ECT four times a week for 3 consecutive weeks
  Arms: ECT treatment
Drug: Drug treatment — Patients only have antipsychotic drugs
  Other Names: olanzapine,clozapine,magnesium valproat,etc.
  Arms: Drug treatment

SUMMARY:
For more severe and treatment-resistant cases in schizophrenia and bipolar disorder, electroconvulsive therapy (ECT) is often very effective. The purpose of this study is to investigate the brain structure and function changes after ECT treatment. The neuroimaging marker which may predict the outcome of ECT is also studied in this research.

ELIGIBILITY:
Inclusion Criteria:

* International classification of diseases (ICD) diagnosis of Schizophrenia and bipolar disorder;
* Ages 15-70
* All participants are ethnic Han
* Not received ECT treatment before
* PANSS ≥ 60 for schizophrenia subjects
* The patient's written informed consent can be obtained. If the patient is incapacitated during the onset period, the written informed consent of the legal guardian is required.

Exclusion Criteria:

* Those with mental retardation, generalized developmental disorders,delirium, dementia, memory impairment or cognitive impairment that meet the diagnostic criteria of ICD-10;
* Patients with cognitive impairment, such as Parkinson's, multiple sclerosis, stroke, and patients who meet the diagnostic criteria for ICD-10 alcohol dependence (except nicotine dependence);
* The course of the disease is very short (fast phase inversion), such as 4 or more different mood abnormalities (depression, mild mania, mania, mental illness) in one year;
* With severe unstable physical diseases; diagnosed diabetes, thyroid disease, hypertension, heart disease, etc.;
* Narrow angle glaucoma;
* With a history of epilepsy, except those with febrile seizures;
* Have or have had drug-induced malignant syndrome and severe tardive dyskinesia;
* With serious suicide attempts;
* Cannot take medication as directed by their doctors, or who do not have guardians;
* Pregnant or lactating women, or those who plan to become pregnant;

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Positive And Negative Syndrome Scale(PANSS)for Schizophrenia; | 3 time points: baseline, the end of the three-week treatment，3 months after ECT or drugs treatment
  Scales changes from baseline will be documented after three weeks treatment and 3 months follow-up visit.
Change of Bech-Rafaelsen Mania Rating Scale (BRMS) for Bipolar disorder | 3 time points: baseline, the end of the three-week treatment，3 months after ECT or drugs treatment
  Scales changes from baseline will be documented after three weeks treatment and 3 months follow-up visit.
Change of Hamilton Anxiety Scale (HAMA) for Bipolar disorder | 3 time points: baseline, the end of the three-week treatment，3 months after ECT or drugs treatment
  Scales changes from baseline will be documented after three weeks treatment and 3 months follow-up visit.
Change of Hamilton depression scale (HAMD) for Bipolar disorder | 3 time points: baseline, the end of the three-week treatment，3 months after ECT or drugs treatment
  Scales changes from baseline will be documented after three weeks treatment and 3 months follow-up visit.

SECONDARY OUTCOMES:
Changes of brain gray matter, white matter and functional based on MRI data analysis | 2 time points:baseline, the end of the three-week treatment]
  The changes of gray matter volume,structural integrity of white matter,and brain function during resting state after treatment will be analyzed.
Change of Mini-Mental State Examination | 3 time points: baseline, the end of the three-week treatment，3 months after ECT or drugs treatment
  Scale change from baseline will be documented after three weeks treatment and 3 months follow-up visit.

IPD SHARING:
Plan to Share IPD: No